CLINICAL TRIAL: NCT01092975
Title: A Phase I Safety Study of Phenylephrine Applied Topically to the Oral Mucosa in Cancer Patients Receiving Radiation to Sub-mandibular Lymph Nodes
Brief Title: Safety of Phenylephrine for Oral Mucositis Prevention
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: formulation/dose changes; planned changes to safety monitoring/reporting
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2009-0077; NCI-2011-00742 (Registry Identifier: NCI Trial ID); CO09901 (Other: UWCCC)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Mucositis; Stomatitis
Keywords: radiotherapy
MeSH Terms: conditions — Mucositis; Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1.25 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 2.5 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 5.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 10.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 20.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 40.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 60.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution
- 80.0 mg phenylephrine (Experimental)
  Interventions: Drug: phenylephrine solution

INTERVENTIONS:
Drug: phenylephrine solution — Subjects will receive up to 40 dose of topical phenylephrine at the specified dose level.

SUMMARY:
The purpose of this study is to determine if applying the drug phenylephrine to the inside of the mouth can be done safely and is tolerable to use in cancer patients receiving radiation to the Sub-mandibular lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients scheduled to receive at least 5 weeks of radiation therapy to the sub-mandibular lymph nodes
* normal ECG
* normal blood pressure

Exclusion Criteria:

* untreated cardiac disease
* connective tissue disorders
* open sores, wound, ulcerations to oral cavity
* allergy to phenylephrine
* know untreated hypertensin
* abnormal ECG in past 6 months
* taking prescription monoamine oxidase inhibitor (MAOI)
* are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety: the presence or absence of mucosal or systemic toxicity related the the topical application of phenylephrine. | 24 months

SECONDARY OUTCOMES:
Efficacy: the the mucositis severity area-under-the-curve (AUC) where the severity of oral mucositis on each treatment day will be scored, summed, and plotted graphically. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James F Cleary, MBBS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/